CLINICAL TRIAL: NCT04521777
Title: Pilot Study Evaluating Changes in Physical Function Measures in Stem Cell Transplant Patients at Risk for Steroid Myopathy
Brief Title: Studying Changes in Physical Function Measures in Stem Cell Transplant Patients at Risk for Steroid Myopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated early due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0141; NCI-2020-05460 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0141 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-11; First posted 2020-08-21 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Acute Graft Versus Host Disease
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (exercise intervention) (Experimental): Patients complete a physical function test over 15 minutes at baseline, and at days 14, 28, and 56. Patients also participate in an 8-week home-based strengthening and walking program consisting of a strengthening/resistance program for 30 minutes, 3 times a week, and walking program for 20-30 minutes at least 3 times a week.
  Interventions: Behavioral: Exercise Intervention; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Participate in an 8-week home-based strengthening and walking program
Other: Physical Performance Testing — Complete a physical function test
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial investigates the changes in physical and functional tests over time in patients with suspected acute graft versus host disease (from a hematologic stem cell transplant) who started treatment with corticosteroids. Sometimes the transplanted cells from a donor can attack the body's normal cells (called graft-versus-host disease). Steroids are used to treat suspected graft-versus-host disease. Steroid myopathy (muscle weakness and fatigue) is a significant side effect of high dose steroid therapy, and can impair activities of daily of life. The goal of this trial is to learn how patients' physical activities and functions change over time while on GVHD-steroid treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform a pilot study to estimate the change in six physical and functional tests over time in patients with suspected acute graft-versus-host disease (GVHD) who have been initiated on treatment with corticosteroids.

SECONDARY OBJECTIVES:

I. To describe and potentially define steroid myopathy by following the patterns of the muscle loss and functional impairment in this population of patients.

II. To follow steroid myopathy and describe its incidence, its severity, and the impact on non-relapse mortality in a homogeneous population of patients with suspected acute graft-versus-host disease (GVHD) who have been initiated on treatment with corticosteroids at a quaternary institution in the inpatient and outpatient setting.

III. To estimate the adherence to an intermittently supervised exercise program in hematopoietic stem cell transplantation (HSCT) patients who are at risk of developing steroid myopathy.

OUTLINE:

Patients complete a physical function test over 15 minutes at baseline, and at days 14, 28, and 56. Patients also participate in an 8-week home-based strengthening and walking program consisting of a strengthening/resistance program for 30 minutes, 3 times a week, and walking program for 20-30 minutes at least 3 times a week.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing and able to give written informed consent and to comply with all of the study visits and procedures
* Age >= 55 years, or with a Sorror co-morbidity index of >= 3
* Post allogenic hematopoietic stem cell transplantation using bone marrow, peripheral blood or cord blood; or after pre planned donor lymphocyte infusion
* Presumptive diagnosis of acute GVHD necessitating high-dose corticosteroid treatment (with an approximate starting dose of methylprednisolone equivalent of 2 mg/kg/day)
* Within 5 days of receiving corticosteroid treatment
* ECOG (Eastern Cooperative Oncology Group) performance status of 0, 1, or 2 or equivalent Karnofsky score of 60 or higher
* The patient is referred to the study by their stem cell transplant attending physician

Exclusion Criteria:

* Non-English speaking
* Underlying unstable cardiac or pulmonary disease in the opinion of the investigator that limits participant involvement in exercise
* Has a pre-transplant echocardiogram with ejection fraction < 45%
* Requires supplemental oxygen to maintain oxygen (O2) saturation > 92%
* Musculoskeletal injury that precludes participation in an exercise program
* Inability to participate in a structured exercise program
* Patients for whom the physician feels is unsafe for an exercise program
* Platelets equal to or less than 10,000 or evidence of active bleeding
* Patients who are unable to understand or follow through with the exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: An T Ngo-Huang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ngo-Huang A, Yadav R, Bansal S, Williams J, Wu J, Fu JB, Alousi AM, Bruera E. An Exploratory Study on Physical Function in Stem Cell Transplant Patients Undergoing Corticosteroid Treatment for Acute Graft-Versus-Host-Disease. Am J Phys Med Rehabil. 2021 Apr 1;100(4):402-406. doi: 10.1097/PHM.0000000000001660. PMID 33278131
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were treated with high dose corticosteroid for Acute Graft Versus Host Disease at MD Anderson Cancer Center between October 2015 and April 2017.
Groups:
- All Participants: In this single-arm trial, patients who were started on high dose corticosteroids (methylprednisolone or equivalent, 2mg/kg/day) for suspected Acute Graft Versus Host Disease were enrolled on the trial. In order monitor for muscle weakness, serial physical function measures were obtained (baseline, Day 14 after enrollment, Day 28, and Day 56). All enrolled patients were also instructed on a home-based exercise program.
Period: Overall Study
Arm/Group | All Participants
Started | 24
Completed | 20
Not Completed | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Data for the 23 participants were analyzed. 1 participant was inevaluable.
Arm/Group | All Participants
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23
Body Mass Index [Median (Full Range); unit: kg/m^2] | 29 [19 to 39]
Primary Cancer [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia | 7
  Myelodysplastic Syndrome | 4
  B cell Lymphoma | 3
  Chronic Myeloid Leukemia | 4
  Chronic Lymphocytic Leukemia | 2
  Acute Lymphocytic Leukemia | 2
  Myelofibrosis | 1
Cancer Status [Count of Participants; unit: Participants]
  Active | 6
  Refractory | 2
  Remission | 15
Graft Source [Count of Participants; unit: Participants]
  Bone marrow | 4
  Peripheral Blood | 19

OUTCOME MEASURES:

1. Primary Outcome: 6 Minutes Walk Test
Description: 6 minute walk test (measured in meters) was conducted on Baseline, Day 14, Day 28 and Day 56 and measured the median changes for Day 14 minus Day 0, Day 28 minus Day 0, and Day 56 minus Day 0.
Time Frame: Baseline, Day 14, Day 28 and Day 56
Measure: Median (Full Range); unit: meters
Arm/Group | All Participants
Number analyzed (Participants) | 23
meters
  Day 14 minus Day 0 | -9.25 [-354 to 174]
  Day 28 minus Day 0 | -20 [-360 to 185]
  Day 56 minus Day 0 | -23 [-360 to 263]

2. Primary Outcome: 5 Times Sit to Stand (5xSTS)
Description: 5xSTS was measured in seconds on Baseline, Day 14, Day 28 and Day 56 and measured the median changes for Day 14 minus Day 0, Day 28 minus Day 0 and Day 56 minus Day 0.
Time Frame: Baseline, Day 14, Day 28 and Day 56
Measure: Median (Full Range); unit: seconds
Arm/Group | All Participants
Number analyzed (Participants) | 23
seconds
  Day 14 minus Day 0 | 1.6 [-11 to 37]
  Day 28 minus Day 0 | 4.0 [-16 to 37]
  Day 56 minus Day 0 | 1.85 [-14.5 to 37]

3. Primary Outcome: Brooke Scale for Myopathy
Description: Brooke Scale for myopathy (a score from 0 to 6, with 6 being the best score with full range of motion of the arms) was measured on Baseline, Day 14, Day 28 and Day 56 and measured the median changes for Day 14 minus Day 0, Day 28 minus Day 0 and Day 56 minus Day 0
Time Frame: Baseline, Day 14, Day 28 and Day 56
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 23
score on a scale
  Day 14 minus Day 0 | 0 [-6 to 0]
  Day 28 minus Day 0 | 0 [-6 to 0]
  Day 56 minus Day 0 | 0 [-6 to 0]

4. Primary Outcome: Modified Adult Myopathy Assessment Tool
Description: The modified Adult Myopathy Assessment Tool assigns a numerical score to a series of physical tasks (arm raise [0 to 3], sustained arm raise [0 to 4], single sit-to-stand [0 to 3], sustained hip flexion [0 to 4], and sustained knee extension [0 to 4]). The total score of all test components (0 to 18) is reported, with 18 as the highest score for muscle function and endurance.
Time Frame: Baseline, Day 14, Day 28 and Day 56
Measure: Median (Full Range); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 23
score on a scale
  Day 14 minus Day 0 | 0 [-18 to 3]
  Day 28 minus Day 0 | -1 [-18 to 3]
  Day 56 minus Day 0 | -3 [-18 to 3]

5. Primary Outcome: Knee Extensors Strength
Description: Knee Extensors Strength (in pounds) was measured on Baseline, Day 14, Day 28 and Day 56 and measured the median change for Day 14 minus Day 0, Day 28 minus Day 0 and Day 56 minus Day 0.
Time Frame: Baseline, Day 14, Day 28 and Day 56
Measure: Median (Full Range); unit: pounds
Arm/Group | All Participants
Number analyzed (Participants) | 23
pounds
  Day 14 minus Day 0 | -6.43 [-32.2 to 14.25]
  Day 28 minus Day 0 | -4.83 [-32.2 to 11.78]
  Day 56 minus Day 0 | -14.30 [-32.2 to 12.73]

6. Primary Outcome: Hip Flexors Strength
Description: Hip Flexors Strength (in pounds) was measured on Baseline, Day 14, Day 28 and Day 56 and measured the median changes for Day 14 minus Day 0, Day 28 minus Day 0 and Day 56 minus Day 0.
Time Frame: Baseline, Day 14, Day 28 and Day 56
Measure: Median (Full Range); unit: pounds
Arm/Group | All Participants
Number analyzed (Participants) | 23
pounds
  Day 14 minus Day 0 | -3.21 [-37.03 to 16.65]
  Day 28 minus Day 0 | -4.98 [-37.03 to 20.65]
  Day 56 minus Day 0 | -4.90 [-37.03 to 20.78]

ADVERSE EVENTS:
Time Frame: 56 Days
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 3/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/77/NCT04521777/Prot_SAP_000.pdf